CLINICAL TRIAL: NCT00666965
Title: A Placebo-Controlled Study for SPM 962 in RLS Patients
Brief Title: A Placebo-Controlled Study for SPM 962 in Restless Legs Syndrome (RLS) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 243-07-003
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Results first posted 2014-04-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-03

CONDITIONS: Idiopathic Restless Legs Syndrome
Keywords: SPM 962; rotigotine; Idiopathic Restless Legs Syndrome; RLS
MeSH Terms: interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): inactive placebo
  Interventions: Drug: SPM 962
- 2 (Experimental): 2.25 mg first week: 2.25 mg 1 sheet plus placebo 1 sheet 2nd to 6th week :2.25mg 1 sheet plus placebo 2 sheets
  Interventions: Drug: SPM 962
- 3 (Experimental): 4.5 mg/body first week : 2.25 mg 2 sheets 2nd to 6th week : 2.25 mg 2 sheets pus placebo 1 sheet
  Interventions: Drug: SPM 962
- 4 (Experimental): 6.75 mg/body first week : 2.25 mg 2 sheets 2nd to 6th week : 2.25 mg 3sheets
  Interventions: Drug: SPM 962

INTERVENTIONS:
Drug: SPM 962 — transdermal application, 1 time per day, 0-6.75 mg/body, titration, 6weeks
  Other Names: rotigotine

SUMMARY:
The primary objective of this study is to investigate efficacy and safety of SPM 962 in Japanese RLS patients in a multi-center, placebo-controlled double-blind parrallel group comparative study following once-daily multiple transdermal doses of SPM 962 within a range of 2.25 to 6.75 mg/day. Recommended maintainance dose range is also to be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 20 and more and less than 80 years of age and is able to think about her/his participation at the time of informed consent.
2. Subject meets the diagnosis of idiopathic RLS based on the 4 cardinal clinical features according to the IRLSSG/NIH.
3. The following subject will be included in the study

   * Subject is not currently receiving treatment for RLS.
   * Subject has previously received treatment of either L-dopa or dopamine agonists and efficacy was observed in either of drugs.
4. At baseline, subject has a score of ≧ 15 on the IRLS sum score and RLS symptoms occur twice and more a week (≧score 2 in IRLS Question 7)
5. Subject has a score of ≧ 4 on the CGI Severity score at baseline

Exclusion Criteria:

1. Subject has secondary RLS in association with renal impairment such as uremia，iron deficiency anemia, and drug associated symptoms.
2. Subject has, is suspected of having or has a history of sleep disorders such as sleep apnea syndrome, narcolepsy, sleep attacks/sudden onset of sleep.
3. Subject has additional clinically relevant concomitant diseases or symptoms such as polyneuropathy (including diabetic neuropathy), akathisia，claudication varicoses，muscle fasciculation，painful legs moving toes and radiculopathy.
4. Subject has other central nervous diseases like Parkinson's disease, dimentia, progressive supranuclear paresis, multisystem atrophy, Huntington's Chorea, amyotrophic lateral sclerosis, or Alzheimer's disease.
5. At screening or baseline, subject has psychiatric condition like confusion, hallucination, delusion, excitation, deliria, abnormal behaviour.
6. Subject has orthostatic hypotension or systolic BP marks ≦ 100 mm Hg and with a decrease of BP from supine to standing position of ≧ 30 mm Hg.
7. Subject has a history of epilepsy, convulsion etc.
8. Subject has serious cardiac dysfunction and/or arrhythmias (e.g., congestive heart failure Class III or IV by NYHA, myocardial infarction, angina pectoris, conduction system dysregulations, second or third degree AV block, complete left bundle branch block, sick-sinus-syndrome, ventricular fibrillation within twelve months prior to enrollment).
9. Subject has arrhythmia and receiving Class Ia antiarrhythmic drugs(e.g., quinidine, procainamide), Class III antiarrhythmic drugs (e.g., amiodarone, sotalol)
10. At screening and baseline, subject develops serious ECG abnormality. Subjects has QTc-interval >450 msec twice at screening. Subject has a the average QTc-interval from two ECGs >450 msec in males and >470 msec in females at baseline.
11. Subject has long QT syndrome congenital.
12. Subject has a serum potassium level < 3.5 mEq/L at screening.
13. Subject has a total bilirubin ≧3.0 mg/dL or AST(GOT) and/or ALT(GPT) greater than 2.5 times the upper limit of the reference range (or ≧100 IU/L) at screening.
14. Subject has BUN ≧ 30 mg/dL or serum creatinine ≧2.0 mg/dl at screening.
15. Subject has a history of allergic reaction to topical agents such as transdermal patch.
16. Subject is pregnant or nursing or woman who plans pregnancy during the trial.
17. Subject pursues shift work or is subject to other continuous non-disease-related life conditions which do not allow regular sleep at night.
18. Subject has autoimmune disease, chronic active hepatitis or immune deficiency disorder.
19. Subject has a malignant neoplastic disease requiring therapy within twelve months prior to screening.

19. Subject received an investigational drug from other clinical trial within the last 12 months prior to baseline.

20. Subject is judged to be inappropriate for this trial by investigator on the other than above.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — New Product Evaluation Development
Locations (8):
- Japan (8):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: placebo transdermal patch
- 2.25 mg/Day: SPM962 maintein dose: 2.25 mg/day
- 4.5 mg/Day: SPM962 maintein dose: 4.5mg/day
- 6.75 mg/Day: SPM962 maintein dose: 6.75 mg/day
Period: Overall Study
Arm/Group | Placebo | 2.25 mg/Day | 4.5 mg/Day | 6.75 mg/Day
Started | 58 | 57 | 58 | 57
Completed | 55 | 53 | 56 | 42
Not Completed | 3 | 4 | 2 | 15
Not completed — Adverse Event | 0 | 2 | 1 | 9
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 2
Not completed — Discontinuation criteria | 2 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: 3 subjects (1 for each placebo, 4.5 mg/day and 6.75 mg/day arm) were excluded by criteria
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 2.25 mg/Day | 4.5 mg/Day | 6.75 mg/Day | Total
Number analyzed (Participants) | 57 | 57 | 57 | 56 | 227
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 48 | 48 | 49 | 48 | 193
  >=65 years | 9 | 9 | 8 | 8 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (13.1) | 50.6 (13.0) | 48.3 (14.1) | 51.0 (12.4) | 49.6 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 41 | 33 | 32 | 143
  Male | 20 | 16 | 24 | 24 | 84
Region of Enrollment [Number; unit: participants]
  Japan | 57 | 57 | 57 | 56 | 227

OUTCOME MEASURES:

1. Primary Outcome: Change of International Restless Legs Syndrome Study Group Rating Scale (IRLS) Score From the Baseline to the End of Titration/Maintenance Period
Description: IRLS is a scale for assessing severity of restless legs syndrome symptoms. IRLS consists of ten questions. Each question is scored from 4 for the first (top) answer (usually 'very severe') to 0 for the last answer (usually none).
  The sum of the score of each question serves as the scale score.
  The scale scoring criteria are: Mild (score 1-10); Moderate (score 11-20); Severe (score 21-30); Very severe (score 31-40). A decrease in the scores means improvement.
Time Frame: Baseline, end of maintenance period at 6 weeks
Population: Full analysis set (FAS), last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | 2.25 mg/Day | 4.5 mg/Day | 6.75 mg/Day
Number analyzed (Participants) | 57 | 55 | 56 | 51
scores on a scale | -9.8 (7.2) | -10.7 (6.3) | -14.4 (7.2) | -14.1 (8.8)

2. Secondary Outcome: Clinical Global Impression (CGI) Severity
Description: CGI is a clinician-reported scale for assessing severity of illness.
  The sale scoring criteria are 1: Normal, not at all ill, 2: Borderline ill, 3: Mildly ill, 4: Moderately ill, 5: Markedly ill, 6: Severely ill, 7: Among the most extremely ill patients.
Time Frame: Baseline, 2 weeks, 4 weeks and 6 weeks. The data at 6 weeks after dosing is shown.
Population: FAS, LOCF
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 2.25 mg/Day | 4.5 mg/Day | 6.75 mg/Day
Number analyzed (Participants) | 57 | 55 | 56 | 51
Percentage of Participants
  Decreased | 73.7 | 83.6 | 92.9 | 86.3
  Increased | 1.8 | 1.8 | 0.0 | 3.9
  Decreased to 1 or 2 | 12.3 | 18.2 | 41.1 | 39.2
  Subjects with CGI score 5 | 8.8 | 12.7 | 3.6 | 7.8
  Subjects without improvement | 26.3 | 16.4 | 7.1 | 13.7
  4 at baseline and stayed at 4 | 26.5 | 13.3 | 10.7 | 10.7
  5 at baseline and decreased to 1 or 2 | 0 | 24.0 | 46.4 | 30.4

3. Secondary Outcome: Patient Global Impression (PGI) Improvement
Description: The PGI-I is a self-rated 7-point scale, with scores ranging from 1 (very much improved) to 7 (very much worse), that assesses the improvement or worsening of a patient's illness relative to baseline at the beginning of the intervention. Scores: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; or 7=very much worse. Moderate and marked improvement = score of 1 or 2, Without improvement = score of 4, Marked and moderate aggravation = score of 6 or 7.
Time Frame: Baseline, 4 weeks and 6 weeks. The data at 6 weeks after dosing is shown.
Population: FAS, LOCF
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 2.25 mg/Day | 4.5 mg/Day | 6.75 mg/Day
Number analyzed (Participants) | 56 | 54 | 56 | 48
Percentage of Participants
  Moderate and marked improvement | 55.4 | 70.4 | 82.1 | 85.4
  Without improvement | 17.9 | 3.7 | 3.6 | 6.3
  Moderate and marked aggravation | 0.0 | 0.0 | 1.8 | 0.0

4. Secondary Outcome: The Pittsburgh Sleep Quality Index (PSQI)
Description: PSQI is a scale for assessing severity of sleep disorders. The score ranges from 0 to 21. 0 indicates "no difficulty" and 21 indicates "severe difficulty". A decrease in the scores means improvement.
  The data at 6 weeks after dosing is shown.
Time Frame: Baseline, every two weeks
Population: FAS, LOCF
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 2.25 mg/Day | 4.5 mg/Day | 6.75 mg/Day
Number analyzed (Participants) | 56 | 54 | 56 | 47
Percentage of Participants
  Subjects with ≥60% decrease | 7.1 | 16.7 | 23.2 | 23.4
  Subjects with ≥50% decrease | 25.0 | 27.8 | 39.3 | 44.7

5. Secondary Outcome: Medical Outcome Study (MOS) Short-Form 36-Item Health Survey (SF-36)
Description: Mean Change from baseline in MOS Short Form SF-36 to 6 weeks after dosing. SF-36 is a scale for assessing health status in clinical practice and research. The scores of 36 questions are summarized into 7 sub-scales. In each sub-scale which range is 0-100, a higher score indicates a better health status. Thus a increase in the scores means improvement.
Time Frame: Baseline, every two weeks
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | 2.25 mg/Day | 4.5 mg/Day | 6.75 mg/Day
Number analyzed (Participants) | 56 | 54 | 56 | 47
Scores on a scale
  Physical functioning | 1.1 (8.1) | 1.6 (9.6) | 2.8 (12.7) | 0.1 (6.1)
  Role physical | -0.4 (18.0) | 1.7 (18.7) | 1.3 (15.8) | 0.9 (11.9)
  Bodily pain | -1.7 (25.0) | 5.0 (28.0) | 1.7 (27.4) | 12.6 (19.7)
  General health | 3.4 (16.4) | 2.5 (10.5) | 4.6 (14.8) | 4.9 (12.9)
  Vitality | 6.3 (16.6) | 6.5 (17.2) | 3.6 (19.9) | 6.5 (18.6)
  Social functioning | -0.2 (19.3) | 4.4 (17.0) | 1.1 (18.4) | 4.0 (12.5)
  Role emotional | -0.1 (18.4) | 5.7 (18.4) | 4.2 (18.7) | 0.7 (16.6)

6. Secondary Outcome: IRLS Each Parameter
Description: IRLS is a scale for assessing severity of restless legs syndrome symptoms. IRLS consists of ten questions. Each question is scored from 4 for the first (top) answer (usually 'very severe') to 0 for the last answer (usually none).
  The sum of the score of each question serves as the scale score. The scale scoring criteria are: Mild (score 1-10); Moderate (score 11-20); Severe (score 21-30); Very severe (score 31-40). A decrease in the scores means improvement.
  The percentage of subjects with -3 or -4 changes from baseline in each parameter at 6 weeks after dosing is shown.
Time Frame: Baseline, every two weeks
Population: FAS, LOCF
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 2.25 mg/Day | 4.5 mg/Day | 6.75 mg/Day
Number analyzed (Participants) | 57 | 55 | 56 | 51
Percentage of Participants
  -4 (RLS discomfort) | 0.0 | 0.0 | 0.0 | 3.9
  -3 (RLS discomfort) | 7.0 | 1.8 | 16.1 | 19.6
  -4 (need to move around due to RLS symptoms) | 0.0 | 0.0 | 3.6 | 2.0
  -3 (need to move around due to RLS symptoms) | 10.5 | 9.1 | 16.1 | 25.5
  -4 (discomfort relief by moving around) | 0.0 | 0.0 | 1.8 | 2.0
  -3 (discomfort relief by moving around) | 7.0 | 9.1 | 26.8 | 13.7
  -4 (severity of RLS as a whole) | 0.0 | 0.0 | 0.0 | 2.0
  -3 (severity of RLS as a whole) | 1.8 | 3.6 | 12.5 | 19.6
  -4 (RLS symptoms frequency) | 1.8 | 3.6 | 3.6 | 9.8
  -3 (RLS symptoms frequency) | 7.0 | 7.3 | 26.8 | 19.6
  -4 (average duration of RLS symptoms) | 0.0 | 0.0 | 0.0 | 0.0
  -3 (average duration of RLS symptoms) | 3.5 | 0.0 | 7.1 | 7.8
  -4 (severity of sleep disturbance) | 0.0 | 0.0 | 1.8 | 2.0
  -3 (severity of sleep disturbance) | 3.5 | 12.7 | 12.5 | 21.6
  -4 (tiredness or sleepiness during the day) | 0.0 | 0.0 | 0.0 | 0.0
  -3 (tiredness or sleepiness during the day) | 1.8 | 7.3 | 5.4 | 11.8
  -4 (severity of impact on daily affaires) | 0.0 | 1.8 | 1.8 | 2.0
  -3 (severity of impact on daily affaires) | 5.3 | 3.6 | 3.6 | 7.8
  -4 (severity of mood disturbance) | 0.0 | 0.0 | 1.8 | 0.0
  -3 (severity of mood disturbance) | 5.3 | 5.5 | 1.8 | 7.8

ADVERSE EVENTS:
Time Frame: 7 weeks
Arm/Group | Placebo | 2.25 mg/Day | 4.5 mg/Day | 6.75 mg/Day
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/57 | 0/58 | 0/57
Other Adverse Events (participants affected / at risk) | 29/58 | 37/57 | 50/58 | 44/57
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=58) | 2.25 mg/Day (N=57) | 4.5 mg/Day (N=58) | 6.75 mg/Day (N=57)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (10) | 19 (19) | 25 (29) | 27 (35)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (6) | 6 (7) | 11 (14)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Stomach Discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Application Site Pruritus (General disorders) | 2 (2) | 8 (8) | 11 (11) | 10 (10)
Application Site Reaction (General disorders) | 5 (5) | 6 (6) | 8 (8) | 7 (8)
Application Site Erythema (General disorders) | 4 (4) | 4 (4) | 7 (7) | 7 (7)
Malaise (General disorders) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
Nasopharyngitis (Infections and infestations) | 14 (17) | 12 (13) | 15 (15) | 14 (18)
Blood Creatine Phosphokinase Increased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 3 (3) | 11 (13) | 5 (6)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 4 (5) | 2 (2)
Somnolence (Psychiatric disorders) | 3 (3) | 6 (6) | 11 (13) | 12 (12)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Menses Irregular (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No